CLINICAL TRIAL: NCT04821505
Title: Stress Reduction and Hypertension Prevention in African Americans
Acronym: Milw2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maharishi International University (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Robert Schneider, MD, Director and Dean, Maharishi International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HL60703-02
Record Dates: First submitted 2021-03-17; First posted 2021-03-29 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: High Blood Pressure
Keywords: Blood pressure; Stress reduction; Meditation; lifestyle modification
MeSH Terms: conditions — Hypertension | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: Meditation (Transcendental Meditation, TM) was employed as a lifestyle modification strategy compared to a health education control with exercise and dietary recommendations but with no stress management component
Who Masked: Investigator, Outcomes Assessor
Masking Description: This is a single-blind randomized controlled trial with all data collection personnel and investigators blinded to subjects' treatment status. The study coordinator does not collect data but receives subjects assigned treatment and then to informs them of their treatment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation (Experimental): The Transcendental Meditation program is described as a simple natural technique practiced for 20 minutes twice daily for deep rest and relaxation. Previous studies have shown its feasibility, validity, and reliability in Blacks at risk for CVD.
  Interventions: Behavioral: Transcendental Meditation
- Health Education (Active Comparator): Health education program matched to the experimental intervention for time, attention, and other non-specific factors.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Health Education — didactic classroom instruction on improving ones lifestyle through healthier diet, exercise and control of substance use.
  Other Names: lifestyle modification
  Arms: Health Education
Behavioral: Transcendental Meditation — TM is described as simple technique practiced 20 minutes twice a day for deep rest and relaxation.
  Other Names: TM technique
  Arms: Meditation

SUMMARY:
There are major health disparities in Blacks associated with high blood pressure (BP) and psychosocial stress. We evaluated the effects of lifestyle modification with meditation in Black adults with high normal and normal blood pressure.

Participants (n=304) were randomized to either the Transcendental Meditation technique or Health Education control in addition to usual care for up to 36 months for BP and secondary outcomes.

DETAILED DESCRIPTION:
Background: Blacks suffer from disparities in hypertension, cardiovascular disease (CVD) and currently, coronavirus-19. These conditions are associated with social determinants of health and psychosocial stress. While previous trials demonstrated stress reduction lowering blood pressure in grade I range in Blacks, there is a paucity of clinical trial data in Blacks with high normal and normal BP.

Objective: This randomized controlled trial was conducted to evaluate the effect of stress reduction with the Transcendental Meditation (TM) technique in Black adults with high normal BP and normal BP using International Society of Hypertension (ISH) definitions.

Methods: A total of 304 Black adults with high normal (130-139/85-89 mm Hg) and normal BP (120-129/80-84 mm Hg) were randomized to either TM or health education (HE) arms. BP was recorded at 3, 6, 9, 12, 24, 30, and 36 months after baseline. Linear mixed model analysis was conducted to compare the BP change between TM and HE participants in the high-normal BP and normal-BP groups. Survival analysis for hypertensive events was conducted.

ELIGIBILITY:
Inclusion Criteria:

* self-identified Black women and men
* no current antihypertensive medications
* high normal BP (130-139 mm Hg and/or DBP 85-89 mm Hg) OR
* normal BP (SBP 120-129 mm Hg and/DBP 80-84 mm Hg)

Exclusion Criteria:

* use of antihypertensive medications within the previous 2 months
* history of CVD, ie, myocardial infarction, angina, peripheral artery disease, heart failure, stroke, or renal failure, diabetes, major psychiatric or substance use disorder other life-threatening illness
* lack of signed a consent form

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 1998-05-01 (Actual); Primary Completion 2004-10-01 (Actual); Study Completion 2005-04-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure | baseline 0 to 36 months after baseline
  Both systolic and diastolic BP are measured using standard clinical trial technique recommended by the American Heart Association (AHA)

SECONDARY OUTCOMES:
Anger | baseline 0 to 36 months after baseline
  Anger is measured using the Spielberger State-Trait scale (24 item, 4 pt likert response scale-'almost never to almost always'). Anger-in, anger-out and anger-total scores were recorded as secondary outcomes because anger has been reported to be associated with the progression of BP
Hypertensive events | baseline 0 to 36 months after baseline
  Hypertensive events were defined as SBP ≥140 and/or DBP ≥90 mm Hg on two successive occasions or first prescribed use of antihypertensive medications.
Heart rate | baseline 0 to 36 months after baseline
  Heart rate (bpm) was measured manually by the technician/nurse who counted the subjects pulse in the right radial artery

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Schneider, M.D., Principal Investigator — Maharishi International University

IPD SHARING:
Plan to Share IPD: No